CLINICAL TRIAL: NCT03140891
Title: Nasal High Frequency Oscillation Ventilation(NHFOV) vs. Nasal Continuous Positive Airway Pressure(NCPAP) as Post-extubation Respiratory Support in Preterm Infants With Respiratory Distress Syndrome:a Randomized Controlled Trial
Brief Title: Nasal High Frequency Oscillation Ventilation(NHFOV) for Respiratory Distress Syndrome
Acronym: NHFOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, Director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHFOV
Record Dates: First submitted 2017-04-17; First posted 2017-05-04 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2017-04

CONDITIONS: Respiratory Distress Syndrome; Preterm Infant
Keywords: preterm infant; respiratory distress syndrome; nasal high frequence oscillation ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHFOV (Experimental): NHFOV is used as the supporting mode after extubation
  Interventions: Device: NHFOV
- NCPAP (Active Comparator): NCPAP is used as the supporting mode after extubation
  Interventions: Device: NCPAP

INTERVENTIONS:
Device: NHFOV — NHFOV is used as the noninvasive mode after extubation
  Arms: NHFOV
Device: NCPAP — NCPAP is used as the noninvasive mode after extubation
  Arms: NCPAP

SUMMARY:
In very preterm infants with severe respiratory distress syndrome(RDS), invasive ventilation(IV) , besides nasal continuous positive airway pressure (NCPAP) and early/selective pulmonary surfactant administration, is one key cornerstone to reduce neonatal mortality. However, IV is related to increased risks of bronchopulmonary dysplasia (BPD) and abnormal developmental outcomes in the survival.Weaning from IV is therefore a key procedure to reducing these risks above, and if extubation does not success, repeated intubation and/or prolonged duration of IV will result in increased medical burden and intubation-associated complications and death. How to minimize the need for endotracheal ventilation and subsequent complications constitutes a challenge for neonatologists.

DETAILED DESCRIPTION:
Early weaning from invasive ventilation and avoiding re-intubation remains a focus. Nowadays, early use of noninvasive respiratory support strategies has been suggested to be the most effective pathway to reduce those risks. NCPAP is a widely used way of noninvasive ventilation strategies in preterm infants. However, there is only 60% success rate in avoiding intubation. Supplying with the combined advantages of HFOV and NCPAP with high CO2 removal, no need for synchronisation, less volume/barotraumas, non-invasion and increased functional residual capacity, nasal high frequency oscillation ventilation (NHFOV) is considered as a strengthened version of NCPAP. Thus, NHFOV may be more effective as post-extubation respiratory support to avoid re-intubation and subsequent complications/sequelae comparing with NCPAP in preterm infants. To date, NHFOV was used increasingly in neonatal intensive care unit (NICU) around the world due to its convenient operation and no consideration of synchronisation, and several small studies have reported the beneficial effects of NHFOV in preterm infants. However, there were rare randomized controlled studies compared NHFOV with NCPAP as post-extubation respiratory support strategies in preterm infants.

The purpose of the present study was to compare NHFOV with NCPAP as post-extubation respiratory support on the need for endotracheal ventilation and subsequent complications in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* The gestational age was less than 37 weeks;
* These neonates were diagnosed with RDS and supported by invasive ventilation with synchronized intermittent mandatory ventilation (SIMV. The diagnosis of RDS was based on clinical manifestations and chest X-ray findings. The clinical signs and symptoms of RDS were respiratory distress, tachypnea, nasal flaring, groan, and cyanosis after birth. The typical X-ray picture of RDS showed a grain shadow, air bronchogram or white lung;
* The neonates were ready to be extubated for the first time and subsequent noninvasive ventilation.

Exclusion Criteria:

* parents' decision not to participate;
* major congenital anomalies;
* died or left the NICU within 24 hour.

Eligibility criteria for extubation:

Besides the improved symptoms, X-rays and sufficient spontaneous breathing efforts, the eligibility criteria for extubation were peak inspiratory pressure (PIP) of 15-20 cm H2O, positive end expiratory pressure (PEEP) of 4-6 cm H2O, respiratory rate of 15 to 30, FiO2 from 0.21 to 0.30, hematocrit more than 35%. and arterialized capillary blood gas analysis need to meet the following criteria: pH>7.20, PaCO2<=55 mmHg.

Ages: 30 Minutes to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
intubation rate | 3 days
  the baby was re-intubated due to respiratory failure
total time of hospitalization | 100 days
  the duration of baby in hospital
bronchopulmonary dysplasia(BPD) | at 28 days after birth or 36 weeks'gestational age or at discharge
  bronchopulmonary dysplasia was diagnosed after extubation BPD was defined according to the National Institutes of Health consensus definition

SECONDARY OUTCOMES:
airleaks | 3 days
  airleaks was diagnosed after extubation
Retinopathy of prematurity | 100 days
  Retinopathy of prematurity was diagnosed after extubation
Neonatal necrotizing enterocolitis | 3 days
  Neonatal necrotizing enterocolitis was diagnosed after extubation
Intraventricular hemorrhage | 3 days
  Intraventricular hemorrhage was diagnosed after extubation
mortality rate | 100 days
  the baby died in hospital
patent ductus arteriosus (PDA) | 100 days
  patent ductus arteriosus (PDA) was diagnosed

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen L, Wang L, Ma J, Feng Z, Li J, Shi Y. Nasal High-Frequency Oscillatory Ventilation in Preterm Infants With Respiratory Distress Syndrome and ARDS After Extubation: A Randomized Controlled Trial. Chest. 2019 Apr;155(4):740-748. doi: 10.1016/j.chest.2019.01.014. PMID 30955572